CLINICAL TRIAL: NCT00294528
Title: Comparing Clinical Outcome of 2 Different Total Knee Prostheses: Nexgen LPS-Flex and AGC
Brief Title: Comparing Clinical Outcome of 2 Different Total Knee Prostheses: Nexgen LPS-Flex Versus AGC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2003-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis, knee; total knee arthroplasty; range of motion; satisfaction
MeSH Terms: conditions — Osteoarthritis, Knee; Personal Satisfaction

INTERVENTIONS:
Device: Nexgen LPS-flex and AGC

SUMMARY:
A randomized blinded study is conducted comparing 2 different knee prostheses. Range of motion (ROM), pain, feel of prosthesis, satisfaction and ability to do daily activities are registered at intervals up to one year postop, where patients are informed on which prosthesis they received.

We want to:

* determine whether an increased ROM is achieved with a high-flex knee compared to a standard knee
* and if so, does it matter

DETAILED DESCRIPTION:
100 patients operated on with unilateral TKR are included and randomized to either prostheses.

Patients operated on with bilateral simultaneous TKR receive one of each prostheses but are blinded to which prosthesis is on which side. They have gait analyses performed preop and at intervals up to one year.

ELIGIBILITY:
Inclusion Criteria:

* age below 75 years and active
* preop ROM at least 120 degress flexion
* BMI below 30
* intact ligaments

Exclusion Criteria:

* below 18 years
* unable to understand language or purpose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-01; Study Completion 2010-01

PRIMARY OUTCOMES:
ROM
Pain
Satisfaction
Feel of prosthesis
Gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Husted, consultant, Principal Investigator — head of arthroplasty section; Kristian Stahl Otte, consultant, Principal Investigator — arthroplasty section; Gitte Holm, RN, Principal Investigator — Head nurse of arthroplasty section; Helle Krogshøj Hansen, RN, Principal Investigator — nurse
Locations (1):
- orthopedic department, section of arthroplasty, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Thomsen MG, Husted H, Otte KS, Holm G, Troelsen A. Do patients care about higher flexion in total knee arthroplasty? A randomized, controlled, double-blinded trial. BMC Musculoskelet Disord. 2013 Apr 8;14:127. doi: 10.1186/1471-2474-14-127. PMID 23565578